CLINICAL TRIAL: NCT04534413
Title: Feasibility of the Ultrasmall Composite Optical Fiberscope System for Lung Cancer Observation
Brief Title: Ex-Vivo COF Study for Lung Cancer Observation
Status: Enrolling by invitation | Type: Observational
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Principal Investigator, Kazuhiro Yasufuku, Dr. Kazuhiro Yasufuku, University Health Network, Toronto
Other Study IDs: 20-5565
Record Dates: First submitted 2020-08-26; First posted 2020-09-01 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: composite optical fiberscope (COF) — Fiber Technology

SUMMARY:
Accessing nodules located in the most outer part of the lung is challenging. Tissue that will be removed from the lung will be used to see if we can reach and see the nodule with a very small camera. This camera that may reach in the smaller and outer airways is called a composite optical fiberscope (COF).

The purpose of this study is to evaluate insertion ability of the COF and visualization of the lung tumor by the COF. In order to do so, we plan to evaluate 50 patient samples from the University Health Network over the span of 2 years.

DETAILED DESCRIPTION:
Peripheral pulmonary lesions (PPLs), which include pulmonary nodules and masses, are a common problem in pulmonology practice. The incidence of PPLs will likely increase given the growing adoption of chest CT screening for lung cancer. There are several guidelines available for management of PPLs. If bronchoscopy is selected as the method of diagnosis, conventional bronchoscopy has been one platform used for decades to diagnose PPLs. However, conventional bronchoscopic techniques have significant limitations and overall low diagnostic yield for most PPLs. As a result, innovative bronchoscopic techniques and technologies have evolved over the last decade to diagnose PPLs more accurately. However, accessing to PPLs located in the most peripheral part is still challenging.

As a new method to diagnose and localize cancers, photodynamic diagnosis (PDD) has been gaining attention. PDD is a new technique where a photosensitizer injected intravenously accumulates in the abnormal lesion, then its fluorescence can be detected by a detector. To conduct PDD for PPLs, we collaboratively developed a parallel-type composite optical fiberscope (COF) with an outer tip diameter of 0.97 mm with OK Fiber Technology (Kyoto, Japan). Its small size and flexibility of the tip enable it to be inserted into animal ultrasmall airways. The outer membrane of the fiberscope is made from polytetrafluoroethylene in the COF's insertable section and is hydrophilic coated, which reduces frictional forces when in the contact with the bronchial wall resulting in smooth insertion of the fiberscope. As the COF has illumination fibers and a laser fiber inside, simultaneous white-light and fluorescence imaging with real-time monitoring can be performed to confirm the tip position of the fiberscope during laser irradiation. In this study, we want to evaluate the COF regarding the quality of white-light images and the accessibility of lung tumors located in the peripheral area of the lung.

ELIGIBILITY:
Inclusion Criteria:

1. Any patients scheduled for lobectomy or anatomical segmental resection for malignant lung tumors.
2. 18 years of age or older.

Exclusion Criteria:

1) Any patients with inability to give informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any patients scheduled for lobectomy or anatomical segmental resection for malignant lung tumors
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2020-08-05 (Actual); Primary Completion 2026-12-05 (Estimated); Study Completion 2026-12-05 (Estimated)

PRIMARY OUTCOMES:
insertion ability of the COF using human ex-vivo lungs | 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- Toronto General Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No